CLINICAL TRIAL: NCT04480086
Title: A Phase 1b Study of Mivebresib Alone or in Combination With Ruxolitinib or Navitoclax in Subjects With Myelofibrosis
Brief Title: Safety and Tolerability Study of Mivebresib Tablet Alone or in Combination With Ruxolitinib Tablet or Navitoclax Tablet in Adult Participants With Myelofibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M20-248; 2020-001226-65 (EudraCT Number)
Record Dates: First submitted 2020-07-20; First posted 2020-07-21 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Myelofibrosis (MF)
Keywords: mivebresib; Navitoclax; Ruxolitinib; ABT-263; Cancer; Myelofibrosis; MF; ABBV-075
MeSH Terms: conditions — Primary Myelofibrosis; Neoplasms | interventions — mivebresib; navitoclax; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Segment A: Mivebresib Dose Identification and Optimization (Experimental): Participants who have been previously treated with Janus Kinase inhibitor(s) (JAKi) and stopped such therapy, will receive different dosing regimens and schedules of mivebresib to identify the safe dosing regimen and schedule.
  Interventions: Drug: Mivebresib
- Segment A: Mivebresib Monotherapy (Experimental): Participants will receive the identified safe dosing regimen of mivebresib as monotherapy.
  Interventions: Drug: Mivebresib
- Segment B: Ruxolitinib + Mivebresib "Add-on" Therapy (Experimental): Participants whose disease (myelofibrosis) is inadequately controlled by ongoing ruxolitinib therapy will receive ruxolitinib and mivebresib as "add-on" therapy.
  Interventions: Drug: Mivebresib; Drug: Ruxolitinib
- Segment C: Mivebresib + Navitoclax (Experimental): Participants who have previously been exposed to JAKi, and stopped such therapy, will receive mivebresib and navitoclax.
  Interventions: Drug: Mivebresib; Drug: Navitoclax
- Segment D: Mivebresib + Ruxolitinib (Experimental): Participants who have never received JAKi will receive mivebresib and ruxolitinib.
  Interventions: Drug: Mivebresib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Mivebresib — Tablet: Oral
Drug: Navitoclax — Tablet; Oral
  Other Names: ABT-263
  Arms: Segment C: Mivebresib + Navitoclax
Drug: Ruxolitinib — Tablet; Oral
  Arms: Segment B: Ruxolitinib + Mivebresib "Add-on" Therapy; Segment D: Mivebresib + Ruxolitinib

SUMMARY:
Myelofibrosis (MF) is a bone marrow illness that affects blood-forming tissues in the body. MF disturbs the body's normal production of blood cells, causing extensive scarring in the bone marrow. This leads to severe anemia, weakness, fatigue, and an enlarged spleen. The purpose of this study is to see how safe and tolerable mivebresib is, when given alone, and in combination with navitoclax or ruxolitinib, for adult participants with MF.

Mivebresib is an investigational drug being developed for the treatment of MF. The study has 4 segments - A, B, C, and D. In Segment A, the safe dosing regimen of mivebresib is identified, and then given alone as monotherapy. In Segment B, C, and D, combination therapies of mivebresib with either ruxolitinib or navitoclax are given. Adult participants with a diagnosis of MF will be enrolled. Around 130 participants will be enrolled in 60 sites worldwide.

In Segment A, participants will receive different doses and schedules of oral mivebresib tablet to identify a safe dosing regimen. Additional participants will be enrolled at the identified monotherapy dosing regimen. In Segment B, participants will receive oral ruxolitinib and mivebresib will be given as "add-on" therapy. In Segment C, participants will receive mivebresib and oral navitoclax. In Segment D, participants will receive mivebresib and ruxolitinib. Participants will receive treatment until disease progression or the participants are not able to tolerate the study drugs.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of treatment will be checked by medical assessments, blood and bone marrow tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory values indicative of adequate bone marrow, renal, and hepatic function meeting protocol criteria
* Completion of the Myelofibrosis System Assessment Form (MFSAF) on at least 4 out of the 7 days prior to Day 1 with at least 2 symptoms with a score >=3 or a total score of >=10.
* Documented diagnosis of intermediate or high-risk primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (PPV-MF) or post-essential thrombocytopenia myelofibrosis (PET-MF) as defined by World Health Organization (WHO).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Intermediate - 2, or High-Risk disease as defined by the Dynamic International Prognostic Scoring System (For Segment A only, Intermediate - 1 with palpable splenomegaly >=5 centimeters [cm] below costal margin are also eligible).
* Splenomegaly defined as spleen palpation measurement >= 5 centimeters (cm) below costal margin or spleen volume >= 450 cubic cms as assessed by Magnetic Resonance Imaging (MRI) or Computed Tomography (CT) scan (for Segments A and c, baseline spleen assessment must be obtained > 7 days after discontinuation of most recent Myelofibrosis (MF) therapy. If possible, this assessment should occur within 10 days of Cycle 1 Day 1).

Segment-Specific Prior Therapy Criteria:

* Segment A:

  --Prior exposure to one or more Janus Kinase Inhibitors (JAKi), the most recent of which was discontinued > 28 days prior to Cycle 1 Day 1.
* Segment B:

  * Currently receiving ruxolitinib; AND
  * Willingness to reduce dose (if on a higher dose); and on a stable dose for 14 days or longer prior to Cycle 1 Day 1; AND
  * At least one of the following criteria (a, b, or c):

    1. >= 24 weeks duration of current ruxolitinib course, with evidence of disease that is resistant, refractory, or has lost response to ruxolitinib monotherapy;
    2. < 24 weeks duration of current ruxolitinib course with documented disease progression as defined by any of the following:

       * Appearance of new splenomegaly that is palpable to at least 5 centimeters (cm) below the left costal margin (LCM), in participants with no evidence of splenomegaly prior to the initiation of ruxolitinib.

         * 100% increase in the palpable distance below the LCM, in participants with measurable spleen distance 5 - 10 cm prior to the initiation of ruxolitinib.
         * 50% increase in the palpable distance below the LCM, in participants with measurable spleen > 10 cm prior to the initiation of ruxolitinib.
       * A spleen volume increase >= 25% (as assessed by MRI or CT) in participants with a spleen volume assessment available prior to the initiation of ruxolitinib.
    3. Prior treatment with ruxolitinib for >= 28 days complicated by any of the following:

       * Development of red blood cell transfusion requirement (at least 2 units/month for 2 months).
       * Grade >= 3 adverse events of neutropenia and/or anemia while on ruxolitinib treatment, with improvement or resolution upon dose reduction.
* Segment C:

  * Prior exposure to one or more JAKi (the most recent of which was discontinued > 28 days prior to Cycle 1 Day 1), and are intolerant, resistant, refractory or lost response to teh JAKi.

Exclusion Criteria:

Segment-Specific Prior Therapy Criteria:

* Segment A:

  --Prior exposure to one or more Bromodomain and Extra Terminal (BET) inhibitors.
* Segment B:

  --Prior exposure to one or more BET inhibitors.
* Segment C:

  --Prior exposure to one or more BET inhibitors and/or any B-Cell Lymphoma 2 (BCL2) and/or B-Cell Lymphoma XL (BCLXL) inhibitor, including navitoclax.
* Segment D:

  * Prior exposure to JAKi and/or any BET inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Up To Approximately 1 year from start of study
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve Spleen Volume Reduction of 35% or Greater (SVR35) | Up To Week 24
  Reduction in spleen volume is measured by magnetic resonance imaging (MRI).
Maximum Observed Plasma Concentration (Cmax) of Mivebresib | Up To Week 12
  Maximum observed plasma concentration (Cmax) of Mivebresib.
Time to Cmax (Tmax) of Mivebresib | Up To Week 12
  The amount of time taken to reach Cmax.
Area Under Concentration vs Time Curve (AUC) of Mivebresib | Up To Week 12
  AUC of Mivebresib will be calculated.
Half-Life (t1/2) of Mivebresib | Up To Week 12
  Half-life of Mivebresib will be calculated.
Accumulation Ratio of Mivebresib | Up To Week 12
  Pharmacokinetic parameters will include accumulation ratio of Mivebresib.
Apparent Clearance (CL/F) of Mivebresib | Up To Week 12
  CL/F of Mivebresib will be calculated.
Apparent Volume of Distribution (Vd/F) of Mivebresib | Up To Week 12
  Vd/F of mivebresib will be calculated.
Percentage of Participants With >= 50% Reduction in Total Symptom Score (TSS) | Week 24
  TSS is assessed using the Myelofibrosis Symptom Assessment Form (MFSAF) v4.0. MFSAF v4.0 measures the burden of myelofibrosis-related symptoms. The symptoms are assessed on a 11-point numeric rating scale (NRS) anchored from 0 (absent) to 10 (worst imaginable).
Objective Response Rate (ORR) | Week 24
  ORR is defined as the sum of rates of complete remission (CR) and partial remission (PR).
Maximum Observed Plasma Concentration (Cmax) of Navitoclax | Up To Week 12
  Maximum Observed Plasma Concentration (Cmax) Of Navitoclax.
Time to Cmax (Tmax) of Navitoclax | Up To Week 12
  The amount of time taken to reach Cmax.
Area Under Concentration vs Time Curve (AUC) of Navitoclax | Up To Week 12
  AUC of Navitoclax will be calculated.
Maximum Observed Plasma Concentration (Cmax) of Ruxolitinib | Up To Week 12
  Maximum Observed Plasma Concentration (Cmax) Of Ruxolitinib.
Time to Cmax (Tmax) of Ruxolitinib | Up To Week 12
  The amount of time taken to reach Cmax.
Area Under Concentration vs Time Curve (AUC) of Ruxolitinib | Up To Week 12
  AUC of Ruxolitinib will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (7):
- United States (4):
  - Stony Brook University Hospital /ID# 222653, Stony Brook, New York
  - UC Health - Cincinnati /ID# 224079, Cincinnati, Ohio
  - Thompson Cancer Survival Ctr /ID# 225802, Knoxville, Tennessee
  - University of Texas MD Anderson Cancer Center /ID# 221652, Houston, Texas
- South Africa (2):
  - Wits Clinical Research , Wits Health Consortium (PTY) Ltd /ID# 222669, Johannesburg, Gauteng
  - Alberts Cellular Therapy /ID# 222667, Pretoria, Gauteng
- Inje University Busan Paik Hospital /ID# 224043, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No